CLINICAL TRIAL: NCT02414334
Title: Immediate Versus Delayed Stereotactic Ablative Radiotherapy (SABR) for Patients With Pulmonary Oligometastases From Colorectal Cancer: SABR SCAN Trial A Randomised Clinical Trial
Brief Title: SABR-SCAN Trial for Pulmonary Oligometastases
Acronym: SABR-SCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT2015-02
Record Dates: First submitted 2015-03-30; First posted 2015-04-10 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Oligometastases
Keywords: Oligometastases; Stereotactic ablative radiotherapy (SABR); Metastatic tumours
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate SABR (Active Comparator): Immediate stereotactic ablative radiotherapy (standard arm)
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR)
- Delayed SABR (Experimental): Delayed stereotactic ablative radiotherapy (delayed= treatment six months after randomisation or at disease progression) (experimental arm)
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy (SABR)

SUMMARY:
Rationale:

SABR (Stereotactic ablative radiotherapy) is one of the standard treatment options besides surgical resection for limited lung metastases (oligometastases) from colorectal cancer. High efficacy in terms of local control of metastatic lesions treated has been shown. Nevertheless, the precise effect of SABR upon progression-free- and overall survival in these patients is unknown. To further evaluate and develop local treatment options in metastatic disease, more information is necessary regarding the impact upon - and the pattern of - disease progression of local treatment options such as SABR.

Objective:

To determine the effect upon progression free survival and upon tumorload relative to baseline, both at one year after randomisation of immediate SABR versus delayed SABR (a scan-and-personalise policy). Secondarily, patterns of progression, patient-reported symptoms and quality of life will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* WHO-Performance status (WHO-PS) 0 - 1
* Patients with 1 to 3 lung metastases between 8 mm and 3 cm each, from colorectal cancer. Resection has been considered at a multidisciplinary conference but was not recommended or has been refused by the patient.
* Possibility to define target lesions that fulfil the following criteria:

  * No lesion larger than 3 cm;
  * Not more than 3 metastases ≥ 8 mm in total (lesions smaller than 8 mm in diameter are NOT counted and will NOT be irradiated);
* No prior radiotherapy (SABR or other) within about 2 cm from target lesions (i.e., the distance between prior planning-target-volume (PTV) to actual intended PTV is more than 2 cm AND dose distribution of former radiation permits SABR).
* Primary tumour has been completely removed surgically.
* Metastases outside target organs (e.g. liver metastases or other) are radically treated locally (resection, radiofrequency ablation (RFA), microwave ablation (MWA), stereotactic radiotherapy, or other). Earlier resected or ablated (SABR, RFA, MWA) metastases to lung, liver, or other organ form no exclusion criterion. Brain metastases should be completely resected or treated with stereotactic radiosurgery. Bone metastases should be resected or treated with high dose radiotherapy (equivalent of > 40 Gy) and be asymptomatic.
* Patients at reproductive potential must agree to practice an effective contraceptive method. Women of childbearing potential must not be pregnant or lactating.
* Proficiency in the Dutch language so that quality-of-life questionnaires can be completed in Dutch and absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Before patient randomisation, informed consent must be given according to International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) of the European Union (EU) in accordance with good clinical practice (GCP), and national/local regulations.

Exclusion Criteria:

* Any clinical symptoms possibly or certainly caused by index lungmetastases
* Physical inability to undergo stereotactic radiotherapy (e.g., serious shoulder stiffness)
* Any uncontrolled malignancy other than index colorectal cancer
* Other malignancy within recent two years, even if completely under control (under control = no evidence of disease)
* Failure to comply with any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 12 months after randomisation

SECONDARY OUTCOMES:
Relative change of tumourload expressed as volume of all tumour at one year divided by volume of all tumour at time of randomisation; | 12 months after randomisation
Time to failure of local strategy (TFLS): failure = death or progressive disease NOT amenable to local treatment | when it occurs
Progression of target lesions as measured by CT | 12 months after randomisation
Health-related quality of life profile | Baseline; 3 months after randomisation and at 6, 9, 12, 15, 18, 21 and 24 months
  Euro-Qol 5 dimensions (EuroQoL-5D); Hospital Anxiety and Depression Scale (HADS); European Organization for Research and Treatment of Cancer quality of life questionnaire - lung cancer module (EORTC-QLQ-LC13)
Progression of lesions other than target lesions as measured by CT | 12 months after randomisation

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands